CLINICAL TRIAL: NCT03690076
Title: Development of the Purification of Human Cardiac Mitochondria, Characterization of These Organelles and Validation of the Model in Acute Endocarditis and Obesity
Brief Title: Human Cardiac Mitochondria in Acute Endocarditis and Obesity
Acronym: MITHOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Université d'Auvergne (Other); Auvergne/Rhône-Alpes area (Unknown); Heart and Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-408
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Endocarditis
Keywords: Heart; Mitochondria; Obesity; Endocarditis
MeSH Terms: conditions — Obesity; Endocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: patients with normal weight (23 < BMI < 27) operated for myocardial revascularization by bypass surgery, without infarction, or for valve pathologies without endocarditis
  Interventions: Other: Endocarditis
- Endocarditis: patients with normal weight (23 < BMI < 27) carriers of endocarditis with surgery indication
  Interventions: Other: Endocarditis
- Obese: obese patients (BMI > 30 with waist to hip ratio > or = 1 in men and 0.85 in women) operated for myocardial revascularization by bypass surgery, without infarction, or for valve pathologies without endocarditis
  Interventions: Other: Obese vs. control

INTERVENTIONS:
Other: Endocarditis — Comparison : Endocarditis vs. control
  Groups: Control; Endocarditis
Other: Obese vs. control — Comparisons : Obese vs. control
  Groups: Obese

SUMMARY:
Data about human cardiac mitochondria are cruelly lacking in the literature. However, damages of the activity of these organelles are often the source of abnormal cardiac function in several pathologies. The purpose of this study is to develop a model of purified human cardiac mitochondria, to verify the purity of these organelles and to validate the authenticity of their function in acute endocarditis and obesity, two situations known to alter their activity. Animal studies have shown that microbial infection reduced mitochondrial metabolism whereas obesity increases it. The investigator's hypotheses are the following: 1) acute endocarditis, a form of cardiac microbial infection, reduces the function of human cardiac mitochondria; 2) obesity (body mass index > 30) activates the metabolism of human cardiac mitochondria.

DETAILED DESCRIPTION:
3 groups of patients:

* Controls: patients with normal weight (23 < BMI < 27) operated for myocardial revascularization by bypass surgery, without infarction, or for valve pathologies without endocarditis
* Endocarditis: patients with normal weight (23 < BMI < 27) carriers of endocarditis with surgery indication
* Obese: obese patients (BMI > 30) operated for myocardial revascularization by bypass surgery, without infarction, or for valve pathologies without endocarditis

Comparisons studied:

* Controls vs. endocarditis
* Controls vs. obese patients

ELIGIBILITY:
Inclusion Criteria:

* For the controls : adult patients with normal body weight (23 < BMI < 27) necessitating a cardiac surgery with sternotomy and extracorporeal circulation for myocardial revascularization or valve replacement
* For endocarditis : adult patients with normal body weight (23 < BMI < 27) and endocarditis of bacterial origin necessitating a cardiac surgery with sternotomy and extracorporeal circulation in order to cure a major valve regurgitation or vegetation with higher size than 15 mm with embolic risk
* For obese patients: adult patients with high body weight (BMI > 30 and waist to hip ration > or = 1 for men and 0.85 for women) necessitating a cardiac surgery with sternotomy and extracorporeal circulation for myocardial revascularization or valve replacement

For all the patients:

* Ability to furnish an enlightened agreement
* Menbership of the French social security insurance

Exclusion Criteria:

* Criteria linked to the surgery:
* Surgery of pressing emergency
* Aortic dissection
* Redux surgery

Criteria linked to the patient:

* Protocol refusal
* Protected adult patients
* Previous psychiatric pathology including known addiction states
* Physical or intellectual inability
* Preexisting pathologies such as respiratory failure
* Cardiac failure (ejection fraction < 30% pulmonary hypertenstion > 80 mmHg); aortic counterpulsation; pre-operatory cardiogenic shock
* Severe acute or chronic renal failure with creatinine clearance < 40 ml/min
* Inherited dyslipidemia
* Previous cardiac or thoracic surgery with pericardium opening
* Severe hepatic failure and severe chronic hepatic pathologies
* Evolving neoplasia
* Patients with long course corticoid treatment and with inflammatory diseases
* Patients with double anti-platelet treatment not stopped 48h before the surgery
* Protected people not involved in the study: pregnant women, nursing women, guardianship, deprived of liberty,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function | at day 1 (Moment of the surgery)
  Measurement of oxidative phosphorylation and reactive oxygen species release in isolated human cardiac mitochondria

SECONDARY OUTCOMES:
walk test | at the moment of inclusion in the study (day (-10-5)) and of the end of hospitalization (day +7+10)
  6-minutes walk test
body composition | 1 day before the surgery
  determination of lean masses by impedance-metry
Electrocardiogram : Detections of the rates in events per min of arrhythmias | at days (-10-5), (+7+10), (+30) and (+90)
  Detections of the rates in events per min of arrhythmias (existence of P wave followed by a QRS complex) and atrio-ventricular blocks in all the patients
Membrane lipid composition | at day 1 (at the day of surgery)
  Fatty acid composition of plasma lipids
Markers of oxidative stress in the plasma | at days (0) and (+30) for the plasma and day (0) for the myocardium
  Markers of the oxidative stress in the plasma (amounts of thiol groups and TBARS, activities of SOD, catalase, glutathione peroxidase, ratio between the amounts of GSH and GSSG) and in the myocardium (whole myocardium: ratio between the activities of aconitase and fumarase, amount of protein carbonylation; isolated mitochondria: amount of nitrosylated proteins)
Concentrations of inflammation cytokines in the plasma | at days (-10-5), (0), (+1), (+2), (+7) and (+90)
  Inflammatory cytokines in the plasma (IL-6, IL-1b, TNF-a, fibrinogen, CRP and pro-calcitonin
Semi-quantitative analysis of the amounts of approximatively 6000 molecules in the plasma by metabolomic and lipidomic techniques | at days (0) and (+30)
  Studies performed in the plasma by a U.S. private society (Metabolon)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | at day (+30)
  Exercise testing
Patient follow-up during the hospital stay | morbi-mortality at day (+90)
  quantity of time (h) spent by the patient during the stay in reanimation
Morbi-mortality | measurement during the post-operative 90 days
  rates of deaths and complications (cardiac, renal, hepatic, etc.) during the 90 days following the surgery for all the patients

CONTACTS AND LOCATIONS:
Overall Officials: Kasra AZARNOUSH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Mourmoura E, Rigaudiere JP, Couturier K, Hininger I, Laillet B, Malpuech-Brugere C, Azarnoush K, Demaison L. Long-term abdominal adiposity activates several parameters of cardiac energy function. J Physiol Biochem. 2016 Sep;72(3):525-37. doi: 10.1007/s13105-015-0427-7. Epub 2015 Aug 10. PMID 26255304